CLINICAL TRIAL: NCT04012060
Title: Patient Reported Health-Related Quality of Life After Limited Access and Conventional Aortic Valve Replacement: Design and Rationale of the LIAR-Trial.
Brief Title: Patient Reported Health-Related Quality of Life After Limited Access and Conventional Aortic Valve Replacement
Acronym: LIAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Idserd Klop, Prinicpal Investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL56311.100.16
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Aortic Valve Stenosis; Limited Access Aortic Valve Replacement; Quality of Life
Keywords: Limited access; Aortic valve replacement; upper hemisternotomy; patient reported outcomes; randomized clinical trial
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to both arms with 80 patients per arm. Patients who are unwilling or unable to participate in the randomized study will be treated via conventional median sternotomy with a sutured aortic valve prosthesis and participate in a prospective registry.
Who Masked: Participant, Care Provider
Masking Description: Patients randomized to either the limited access or conventional aortic valve replacement will be blinded for the treatment until day four postoperatively. The patients participating in the prospective registry will not be blinded for their treatment.
  All nurses on the postoperative ward are blinded for the treatment the patients received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional group (Active Comparator): All patients undergoing aortic valve replacement through full sternotomy.
  Interventions: Procedure: Conventional aortic valve replacement
- Limited access group (Experimental): All patients undergoing aortic valve replacement through partial upper hemisternotomy.
  Interventions: Procedure: Limited access aortic valve replacement.
- Registry group (Other): All patients unwilling or unable to participate in the randomized part of the trial.
  All patients will undergo aortic valve replacement through median full sternotomy.
  Interventions: Procedure: Conventional aortic valve replacement

INTERVENTIONS:
Procedure: Limited access aortic valve replacement. — Limited access aortic valve replacement through partial upper hemisternotomy
  Arms: Limited access group
Procedure: Conventional aortic valve replacement — Aortic valve replacement through full median sternotomy
  Arms: Conventional group; Registry group

SUMMARY:
The LIAR-Trial is a single-center, single blind randomized controlled clinical trial comparing patients undergoing isolated AVR via J-shaped upper hemi-sternotomy (UHS) and conventional AVR through a full median sternotomy (FMS). Primary outcome is cardiac-specific quality of life, measured by two domains of the Kansas City Cardiomyopathy Questionnaire (KCCQ), up to one year after surgery.

DETAILED DESCRIPTION:
The LIAR-Trial is a single-center, single blind randomized controlled clinical trial comparing patients undergoing isolated AVR via J-shaped upper hemi-sternotomy (UHS) and conventional AVR through a full median sternotomy (FMS). To reduce potential confounding by differences in implanted valve prostheses, in both arms of the trail, the diseased native aortic valve is planned to be replaced with a rapid deployment stented aortic bioprosthesis (Edwards Intuity Elite Valve System®, Edwards Lifesciences Corporation), the preferred type of valve prosthesis for a limited access approach. Patients will be randomized 1:1 to both arms with 80 patients per arm. Patients who are unwilling or unable to participate in the randomized study will be treated via conventional median sternotomy with a sutured aortic valve prosthesis and participate in a prospective registry.

Primary outcome is cardiac-specific quality of life, measured by two domains of the Kansas City Cardiomyopathy Questionnaire (KCCQ), up to one year after surgery. Secondary outcomes include, but are not limited to: generic quality of life measured with the Short Form-36 (SF-36), postoperative pain, perioperative outcome (i.e. technical success rate, operating time) and postoperative outcome (i.e. 30 day and one-year mortality, complication rate, hospital length of stay, reoperation rate and readmission rate). Questionnaires are administered face to face or by telephone prior to surgery and at one, three, six and twelve months after surgery. In the prospective registry the quality of life questionnaires and all clinical data from the patients will be collected and analyzed the exact same way as the data from patients included and randomized in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an isolated biological aortic valve replacement for a severe and/or symptomatic aortic valve stenosis, defined as:

  * An aortic valve area of ≤1.0cm2, and;
  * Mean valve gradient ≥40mmHg, and/or;
  * A peak velocity of at least 4.0m/s.
* Able to understand the nature of the study and what will be required of them;
* All adult men and non-pregnant women;
* BMI between 18-35.

Exclusion Criteria:

* Inability to give written informed consent;
* Inability to adequately answer the questionnaires;
* Patients requiring additional cardiac surgery during the same procedure;
* Patients requiring a reoperation;
* (relative) contraindications for a limited access approach;
* Undergoing an emergency operation;
* Recent myocardial infarction (<90 days);
* Recent stroke or transient ischemic attack (<6 months);

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac-specific quality of life after aortic valve replacement. | One, three, six and twelve months after surgery
  Change in cardiac specific quality of life after aortic valve replacement measured by the physical limitations and symptoms domains from the Kansas City Cardiomyopathy Questionnaire (KCCQ).

SECONDARY OUTCOMES:
Changes in the self-efficacy domain of the Kansas City Cardiomyopathy Questionnaire (KCCQ) | One, three, six and twelve months after surgery
  Changes in the self-efficacy domain of the KCCQ, after aortic valve replacement.
Changes in social interference domain of the Kansas City Cardiomyopathy Questionnaire (KCCQ) | One, three, six and twelve months after surgery
  Changes in social interference domain of the KCCQ, after aortic valve replacement.
Changes in quality of life domains of the Kansas City Cardiomyopathy Questionnaire (KCCQ) | One, three, six and twelve months after surgery
  Changes in quality of life domain of the KCCQ, after aortic valve replacement.
Change is generic quality of life, assessed with the Physical Component Summary (PCS) of the Short Form-36 (SF-36). | One, three, six and twelve months after surgery
  The SF-36 consists of eight domains: physical functioning, role physical functioning, role emotional functioning, bodily pain, vitality, mental health, role social functioning and general health. These domains can be combined into the PCS and MCS.
Change is generic quality of life, assessed with the Mental Component Summary (MCS) of the Short Form-36 (SF-36). | One, three, six and twelve months after surgery
  The SF-36 consists of eight domains: physical functioning, role physical functioning, role emotional functioning, bodily pain, vitality, mental health, role social functioning and general health. These domains can be combined into the PCS and MCS.
Postoperative sternal pain | First seven days after surgery and one, three, six and twelve months after surgery
  Assessed with a visual analogue score. The VAS is depicted as a straight line from left to right and ranges from 0 (no pain) to 100 (worst imaginable pain)
Perioperative outcomes | During surgery
  aortic cross clamp time (minutes), cardio-pulmonary bypass time (minutes), operating time (minutes) are the main focus. All three outcomes will be measured in minutes.
Clinical outcomes | Up to one year postoperatively.
  30-day mortality and one year mortality rate, complication rate, reoperation rate and readmission rate
Technicall success rate of the aortic valve replacement. | During surgery (peri-operatively)
  Technical success rate is defined as a limited access approach without conversion and placement of the rapid deployment bioprosthesis
Hospital length of stay | Up to one year postoperatively
  The number of days a patient is admitted in the hospital after surgery (aortic valve replacement)
Intensive Care length of stay | Up to one year postoperatively
  The hours a patient has to stay in the Intensive Care Unit postoperatively
Effective orifice area of the aortic valve prosthesis | Up to one year postoperatively
  Postoperatively hemodynamic outcomes of the aortic valve prosthesis that is placed during surgery will be measured. A transthoracic echocardiography will be made during follow-up. The effective orifice area, in square centimeters (cm^2), will be measured.
Need of analgetic drugs | Up to one year postoperatively
  The intake of analgesic drugs (paracetamol and morfine) will be measured.
Mean pressure gradient of the aortic valve prosthesis. | Up to one year postoperatively
  Postoperatively hemodynamic outcomes of the aortic valve prosthesis that is placed during surgery will be measured. A transthoracic echocardiography will be made during follow-up. The mean pressure gradients in milimeters of mercury (mmHg) will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirmani BH, Jones SG, Muir A, Malaisrie SC, Chung DA, Williams RJ, Akowuah E. Limited versus full sternotomy for aortic valve replacement. Cochrane Database Syst Rev. 2023 Dec 6;12(12):CD011793. doi: 10.1002/14651858.CD011793.pub3. PMID 38054555
- [Derived] Klop IDG, van Putte BP, Kloppenburg GTL, Sprangers MAG, Nieuwkerk PT, Klein P. Comparing quality of life and postoperative pain after limited access and conventional aortic valve replacement: Design and rationale of the LImited access aortic valve replacement (LIAR) trial. Contemp Clin Trials Commun. 2021 Jan 12;21:100700. doi: 10.1016/j.conctc.2021.100700. eCollection 2021 Mar. PMID 33506139